CLINICAL TRIAL: NCT05972993
Title: Exploratory, First Time in Human (FTIH), Observer-blind, Randomized, Controlled Study to Evaluate Safety, Reactogenicity and Immunogenicity of Various Doses of GlaxoSmithKline Biologicals SA's (GSK) Investigational Omicron Variant S Glycoprotein (mRNA-CR-04) Vaccine When Administered Intramuscularly in Healthy Adults 18 to 49 Years of Age
Brief Title: A Safety and Immune Response Study to Evaluate Varying Doses of an mRNA Vaccine Against Coronavirus Disease 2019 (COVID-19) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 219112
Record Dates: First submitted 2023-08-01; First posted 2023-08-02 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Master Protocol; Omicron; mRNA
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Dose escalation with sentinel dosing.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Data will be collected in an observer-blind manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Part A, Group 1: mRNA CR-04 10 µg (Experimental): Participants received mRNA 10 micrograms (µg) administered on Day 1.
  Interventions: Biological: mRNA-CR-04 vaccine 10μg
- Part A, Group 1: Placebo (Placebo Comparator): Participants received placebo dose administered on Day 1.
  Interventions: Drug: Placebo
- Part A, Group 2: mRNA CR-04 30 µg (Experimental): Participants received placebo dose administered on Day 1.
  Interventions: Biological: mRNA-CR-04 vaccine 30μg
- Part A, Group 2: Placebo (Placebo Comparator): Participants received placebo dose administered on Day 1.
  Interventions: Drug: Placebo
- Part A, Group 3: mRNA CR-04 100 µg (Experimental): Participants received mRNA 100 µg administered on Day 1
  Interventions: Biological: mRNA-CR-04 vaccine 100μg
- Part A, Group 3: Placebo (Placebo Comparator): Participants received placebo dose administered on Day 1.
  Interventions: Drug: Placebo
- Part B: mRNA CR-04 3 µg (Experimental): Participants received mRNA 3 µg administered on Day 1.
  Interventions: Biological: mRNA-CR-04 vaccine 3μg
- Part B: mRNA CR-04 10 µg (Experimental): Participants received mRNA 10 µg administered on Day 1.
  Interventions: Biological: mRNA-CR-04 vaccine 10μg
- Part B: Placebo (Placebo Comparator): Participants received placebo dose administered on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: mRNA-CR-04 vaccine 10μg — mRNA CR-04 vaccine, 10 µg, is administered intramuscularly into the deltoid muscle of the non-dominant arm on day 1.
  Arms: Part A, Group 1: mRNA CR-04 10 µg; Part B: mRNA CR-04 10 µg
Biological: mRNA-CR-04 vaccine 30μg — mRNA CR-04 vaccine, 30 µg, is administered intramuscularly into the deltoid muscle of the non-dominant arm on day 1.
  Arms: Part A, Group 2: mRNA CR-04 30 µg
Biological: mRNA-CR-04 vaccine 100μg — mRNA CR-04 vaccine, 100 µg, is administered intramuscularly into the deltoid muscle of the non-dominant arm on day 1.
  Arms: Part A, Group 3: mRNA CR-04 100 µg
Drug: Placebo — Placebo is administered intramuscularly into the deltoid muscle of the non-dominant arm on day 1.
  Arms: Part A, Group 1: Placebo; Part A, Group 2: Placebo; Part A, Group 3: Placebo; Part B: Placebo
Biological: mRNA-CR-04 vaccine 3μg — mRNA CR-04 vaccine, 3 µg, is administered intramuscularly into the deltoid muscle of the non-dominant arm on day 1.
  Arms: Part B: mRNA CR-04 3 µg

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immune responses of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) mRNA-CR-04 vaccine construct when administered in healthy adults previously vaccinated with SARS-CoV-2 mRNA vaccines.

DETAILED DESCRIPTION:
There will be dose-escalation in part A of the study with sentinel dosing strategy implemented in each of 3 dosing levels (Group 1; 2; 3). At start, enrollment in Group 1 and 2 will occur simultaneously with the enrolment of 1st participant in Group 1. Each group will consist of 8 sentinel participants, with 6 receiving the mRNA-CR-04 vaccine and 2 receiving a placebo. The safety data from the sentinel participants in both groups, up to Day 8 post-vaccination, will be reviewed by the Internal Safety Review Committee (iSRC).

If no safety signal is observed, vaccination of the non-sentinel participants in that group will continue. If there are no safety signals observed from the sentinel participants in Group 1 and Group 2, the enrollment and vaccination of the sentinel participants in Group 3 will begin.

Part B of the study will commence only after all Part A participants have completed their Day 15 study visits and the Day 15 interim analysis is completed. In Part B, 2 doses of the mRNA-CR-04 vaccine will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Written or witnessed informed consent obtained from the participant prior to performance of any study-specific procedure.
2. Participants, who in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary and study procedures).
3. Has received 2 doses of primary series and booster dose(s) of an authorized or licensed mRNA COVID-19 vaccine (only Moderna or Pfizer vaccines) with the last booster dose administered between at least 6 and 18 months or more prior to screening and has provided documentation of receiving the vaccination series (e.g., vaccination card).
4. Negative for SARS-CoV-2 infection by RT-PCR test at screening within 7 days prior to study vaccination.
5. Is a male or nonpregnant female of 18 to 49 years, inclusive, at screening.
6. If the participant is a woman of childbearing potential (WOCBP), the participant agrees to practice true abstinence or use at least 1 highly effective form of contraception for at least 30 days prior to study vaccination up to 1 month after study vaccination.
7. Agrees to refrain from blood or plasma donation from screening and up to 6 months after vaccination.
8. Is healthy or medically stable as determined by investigator judgment based on medical history, clinical laboratory tests, vital sign measurements, and physical examination findings.

Exclusion Criteria:

1. Has a new onset, clinically significant, abnormal biochemistry or hematology finding [defined as greater than or equal to (>=) Grade 1] at screening (participants with Grade 1 laboratory abnormalities that have been stable for at least 6 months before enrollment may be included in the study).
2. Has any medical disease or condition that, in the opinion of the investigator, precludes study participation. This includes any acute, subacute, intermittent, or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of the trial.
3. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
4. History of myocarditis, pericarditis, second- and third-degree heart block or idiopathic cardiomyopathy, or presence of any medical condition that increases risk of myocarditis or pericarditis, including cocaine abuse, cardiomyopathy, endomyocardial fibrosis, hypereosinophilic syndrome, hypersensitivity myocarditis eosinophilic granulomatosis with polyangiitis, persistent myocardial viral infection (e.g., due to enterovirus or adenovirus).
5. Has an acute febrile illness with a temperature >=38.0 degree Celsius (°C) or >=100.4 degree Fahrenheit (°F) observed by the participant or at the study site within 72 hours prior to study vaccination. Participants with suspected COVID-19 symptoms should be excluded and referred for medical care.
6. Has a history of hypersensitivity or severe allergic reaction, including anaphylaxis, generalized urticaria, angioedema, and other significant reactions to any previous vaccine, or any component of the study vaccine.
7. Has a body mass index greater than (>) 40 Kilograms meter per square (kg/m^2).
8. Has had known close contact with anyone who had a confirmed SARS-CoV-2 infection within 14 days before study vaccination.
9. Has a history of documented SARS-CoV-2 infection or COVID-19 within 6 months before the date of screening visit.
10. Has any self-reported or medically documented clinically significant medical or psychiatric condition. Significant medical conditions include, but are not limited to, the following:

    1. Moderate or severe respiratory disease (e.g., chronic obstructive pulmonary disease, asthma).
    2. Uncontrolled hypertension, defined as an average systolic blood pressure >= 140 millimeters of mercury (mmHg) or an average diastolic blood pressure >= 90 mmHg, based on an average of up to 3 blood pressure measurements.
    3. Clinically significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease).
    4. Neurological or neurodevelopmental conditions (e.g., Down syndrome, dementia, chronic migraine not controlled by medication, epilepsy, stroke or seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain- Barré syndrome, encephalomyelitis, or transverse myelitis).
    5. Ongoing malignancy or recent diagnosis of malignancy in the last 5 years (excluding basal cell and squamous cell carcinoma of the skin).
    6. Tuberculosis or non-tuberculosis mycobacterial infection.
    7. Autoimmune disease, including hypothyroidism without a defined nonautoimmune cause.
    8. Immunodeficiency of any cause, including from solid organ transplant, blood, or bone marrow transplant, or use of other immune-weakening medicine.
    9. Type 1 or 2 diabetes mellitus regardless of disease control.
11. Has any of the following self-reported or medically documented risk factors for severe COVID-19:

    1. Chronic kidney disease
    2. Cerebrovascular disease
    3. Cystic fibrosis
    4. Chronic liver disease
    5. Pulmonary fibrosis
12. Has participated or plans to participate in another investigational study involving any investigational drug or device within 60 days or 5 half-lives, whichever is longer, before study vaccination and throughout the study.
13. Has received a licensed or authorized non-mRNA COVID-19 vaccine (primary series or booster dose).
14. Has received or plans to receive any licensed vaccine within 4 weeks before or after study vaccination. Inactivated vaccines for influenza are permitted during the study if they are administered at least 14 days before or after study vaccination.
15. Is planning to receive an authorized or licensed COVID-19 booster vaccination for the duration of the study (for participants who are not covered by local recommendations to receive booster per current standard of care) OR is planning to receive an authorized or licensed COVID-19 booster vaccination on or before Day 31 of the study (for participants covered by local recommendations to receive booster).
16. Has received or plans to receive immunoglobulins or any blood or blood products within 90 days before study vaccination and throughout the study.
17. Reports chronic use (more than 14 continuous days) of any medication that may be associated with changes in immune function including, but not limited to, systemic corticosteroids exceeding 20 mg/day of prednisone equivalent, allergy injections, immunoglobulins, interferons, immunomodulators, cytotoxic drugs, or other similar or toxic drugs within 6 months of study vaccination. Note: The use of low-dose topical, ophthalmic, inhaled, intra-articular and intranasal steroid preparations is permitted.
18. Pregnant or lactating female.
19. Female participant planning to become pregnant or planning to discontinue contraceptive precautions within 1 month following study vaccination.
20. Participant is an employee or family member of the investigator or study site personnel.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer tohttps://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Group 2: mRNA CR-04 30 µg: Participants received mRNA 30 µg administered on Day 1.
Period: Overall Study
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Started | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6
Completed | 16 | 6 | 17 | 6 | 18 | 6 | 18 | 16 | 6
Not Completed | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo | Total
Number analyzed (Participants) | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.9 (9.8) | 40.2 (8.3) | 39.2 (7.9) | 35.8 (7.0) | 34.7 (8.0) | 37.2 (8.8) | 35.7 (10.5) | 37.7 (7.9) | 41.5 (7.7) | 37.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 10 | 4 | 12 | 4 | 8 | 10 | 3 | 64
  Male | 8 | 3 | 8 | 2 | 6 | 2 | 10 | 8 | 3 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The "All Other Races" category (i.e., ASIAN, BLACK OR AFRICAN AMERICAN, NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER, and WHITE, where 0<n<11) are combined into one category to maintain participant confidentiality and privacy.
  Participants
    All Other Races | 17 | 5 | 18 | 5 | 17 | 6 | 17 | 18 | 5 | 108
    Not reported | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Solicited Administration Site Events
Description: The solicited administration site events are pain, redness, swelling and lymphadenopathy (axillary swelling/ tenderness on the same side of the body as the site of injection). Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 7
Population: Analysis was performed on Solicited Safety Set (SSS) which includes all participants who received at least one dose of investigational products and had solicited events data at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 18 | 18 | 6
Participants
  Pain at administration site | 8 | 0 | 10 | 1 | 15 | 0 | 9 | 6 | 1
  Redness at administration site | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
  Swelling at administration site | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
  Lymphadenopathy | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 3 | 0

2. Primary Outcome: Number of Participants With Any Solicited Systemic Events
Description: The solicited systemic events are fever, headache, myalgia (muscle pain), arthralgia (joint pain), fatigue (tiredness), chills, abdominal pain, vomiting and diarrhea. Fever is defined as body temperature ≥38ºC; preferred location for measuring the temperature is oral. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 7
Population: Analysis was performed on SSS which includes all participants who received at least one dose of investigational products and had solicited events data at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 18 | 18 | 6
Participants
  Fever | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Headache | 5 | 1 | 4 | 1 | 8 | 2 | 6 | 4 | 2
  Myalgia | 4 | 0 | 4 | 2 | 11 | 0 | 6 | 8 | 0
  Arthralgia | 1 | 0 | 3 | 0 | 2 | 1 | 1 | 2 | 0
  Fatigue | 8 | 1 | 7 | 1 | 8 | 2 | 7 | 5 | 1
  Chills | 2 | 0 | 3 | 0 | 3 | 1 | 0 | 2 | 1
  Abdominal Pain | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0
  Vomiting | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  Diarrhea | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1

3. Primary Outcome: Number of Participants With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is an AE that is either not included in the list of solicited events or can be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs include both serious and nonserious AEs. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 30
Population: Analysis was performed on Exposed set, which included all participants who received the dose of the investigational products.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6
Participants | 6 | 0 | 5 | 0 | 4 | 3 | 8 | 2 | 1

4. Primary Outcome: Number of Participants With Any Hematological and Biochemical Laboratory Abnormalities
Description: The hematological and biochemical parameters included alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST), total bilirubin, creatinine, direct bilirubin, basophils, eosinophils increase, erytrocytes, hemoglobin decrease, lymphocytes decrease, mean corpuscular hemoglobin, mean corpuscular volume, monocytes, neutrophils decrease, platelets decrease, white blood cells (WBC) increase. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: Day 1 to Day 15
Population: Analysis was performed on Exposed set. Only participants with data available at specified timepoints were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 18 | 18 | 6
Participants
  ALT: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 17 | 18 | 6
  ALT: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
  ALT: Within (Baseline) - Below (Day 15) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
  ALT: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT: Below (Baseline) - Within (Day 15) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
  ALT: Within (Baseline) - Within (Day 15) | 10 | 4 | 13 | 3 | 14 | 4 | 14 | 14 | 4
  ALT: Above (Baseline) - Within (Day 15) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
  ALT: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT: Within (Baseline) - Above (Day 15) | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0
  ALT: Above (Baseline) - Above (Day 15) | 3 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1
  ALP: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ALP: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: Below (Baseline) - Within (Day 15) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: Within (Baseline) - Within (Day 15) | 16 | 6 | 14 | 6 | 18 | 6 | 17 | 18 | 6
  ALP: Above (Baseline) - Within (Day 15) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: Within (Baseline) - Above (Day 15) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: Above (Baseline) - Above (Day 15) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within (Baseline) - Within (Day 15) | 17 | 5 | 17 | 5 | 16 | 6 | 17 | 18 | 6
  AST: Above (Baseline) - Within (Day 15) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
  AST: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: Within (Baseline) - Above (Day 15) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  AST: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin: Within (Baseline) - Within (Day 15) | 18 | 6 | 17 | 6 | 17 | 6 | 18 | 18 | 6
  Total Bilirubin: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin: Within (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Total Bilirubin: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (Baseline) - Within (Day 15) | 18 | 6 | 16 | 6 | 17 | 5 | 17 | 18 | 5
  Creatinine: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine: Above (Baseline) - Above (Day 15) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Direct Bilirubin: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin: Within (Baseline) - Within (Day 15) | 18 | 6 | 17 | 6 | 18 | 6 | 18 | 18 | 6
  Direct Bilirubin: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin: Within (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Basophils: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within (Baseline) - Within (Day 15) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Basophils: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Within (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils Increase: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Eosinophils Increase: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils Increase: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils Increase: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils Increase: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils Increase: Within (Baseline) - Within (Day 15) | 18 | 6 | 17 | 6 | 17 | 6 | 16 | 17 | 6
  Eosinophils Increase: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils Increase: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils Increase: Within (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils Increase: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Erythrocytes: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Erythrocytes: Below (Baseline) - Below (Day 15) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Erythrocytes: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Erythrocytes: Within (Baseline) - Within (Day 15) | 17 | 5 | 16 | 6 | 18 | 6 | 14 | 16 | 4
  Erythrocytes: Above (Baseline) - Within (Day 15) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Within (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Decrease: number analyzed (Participants) | 18 | 6 | 15 | 6 | 18 | 6 | 16 | 16 | 6
  Hemoglobin Decrease: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Decrease: Within (Baseline) - Below (Day 15) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Decrease: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Decrease: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Decrease: Within (Baseline) - Within (Day 15) | 16 | 6 | 13 | 5 | 18 | 6 | 16 | 16 | 6
  Hemoglobin Decrease: Above (Baseline) - Within (Day 15) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Decrease: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Decrease: Within (Baseline) - Above (Day 15) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Decrease: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Decrease: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Lymphocytes Decrease: Below (Baseline) - Below (Day 15) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Decrease: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Decrease: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Decrease: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Decrease: Within (Baseline) - Within (Day 15) | 17 | 6 | 16 | 5 | 17 | 6 | 16 | 16 | 6
  Lymphocytes Decrease: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Lymphocytes Decrease: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Decrease: Within (Baseline) - Above (Day 15) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Lymphocytes Decrease: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Hemoglobin: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Mean Corpuscular Hemoglobin: Below (Baseline) - Below (Day 15) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Mean Corpuscular Hemoglobin: Within (Baseline) - Below (Day 15) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Hemoglobin: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Hemoglobin: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Hemoglobin: Within (Baseline) - Within (Day 15) | 15 | 6 | 15 | 6 | 18 | 6 | 16 | 16 | 6
  Mean Corpuscular Hemoglobin: Above (Baseline) - Within (Day 15) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Hemoglobin: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Hemoglobin: Within (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Hemoglobin: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Volume: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Mean Corpuscular Volume: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Mean Corpuscular Volume: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Volume: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Volume: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Volume: Within (Baseline) - Within (Day 15) | 12 | 6 | 15 | 6 | 16 | 5 | 15 | 16 | 6
  Mean Corpuscular Volume: Above (Baseline) - Within (Day 15) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Mean Corpuscular Volume: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Volume: Within (Baseline) - Above (Day 15) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Mean Corpuscular Volume: Above (Baseline) - Above (Day 15) | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
  Monocytes: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Monocytes: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (Baseline) - Within (Day 15) | 18 | 6 | 16 | 6 | 18 | 6 | 16 | 17 | 6
  Monocytes: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (Baseline) - Above (Day 15) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Decrease: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Neutrophils Decrease: Below (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Decrease: Within (Baseline) - Below (Day 15) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils Decrease: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Decrease: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Neutrophils Decrease: Within (Baseline) - Within (Day 15) | 14 | 5 | 16 | 6 | 17 | 6 | 15 | 17 | 6
  Neutrophils Decrease: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Decrease: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Decrease: Within (Baseline) - Above (Day 15) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Decrease: Above (Baseline) - Above (Day 15) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decrease: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  Platelets Decrease: Below (Baseline) - Below (Day 15) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decrease: Within (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decrease: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decrease: Below (Baseline) - Within (Day 15) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decrease: Within (Baseline) - Within (Day 15) | 14 | 6 | 16 | 5 | 15 | 5 | 16 | 15 | 6
  Platelets Decrease: Above (Baseline) - Within (Day 15) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Platelets Decrease: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decrease: Within (Baseline) - Above (Day 15) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Platelets Decrease: Above (Baseline) - Above (Day 15) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  WBC Increase: number analyzed (Participants) | 18 | 6 | 17 | 6 | 18 | 6 | 16 | 17 | 6
  WBC Increase: Below (Baseline) - Below (Day 15) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC Increase: Within (Baseline) - Below (Day 15) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  WBC Increase: Above (Baseline) - Below (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC Increase: Below (Baseline) - Within (Day 15) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  WBC Increase: Within (Baseline) - Within (Day 15) | 15 | 5 | 15 | 6 | 16 | 6 | 16 | 17 | 6
  WBC Increase: Above (Baseline) - Within (Day 15) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  WBC Increase: Below (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC Increase: Within (Baseline) - Above (Day 15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC Increase: Above (Baseline) - Above (Day 15) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Any Medically Attended Adverse Events (MAAEs)
Description: A MAAE is an AE for which the participant received medical attention including any symptom or illness requiring hospitalization, or an emergency room visit, or visit to/by a healthcare professional. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 31
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6
Participants | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0

6. Primary Outcome: Number of Participants With Any Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, abnormal pregnancy outcome or any other situation as determined by the investigator. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 31
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Any Adverse Events of Special Interest (AESIs)
Description: AESIs include potential immune-mediated diseases (pIMDs) which are autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology, myocarditis, and pericarditis, virologically confirmed COVID-19 cases, anaphylaxis, or severe hypersensitivity within 24 hours after study investigational product administration. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 31
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Any MAAEs
Description: as for outcome 5
Time Frame: Throughout the study period (Day 1 to Month 6)
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6
Participants | 3 | 1 | 2 | 0 | 3 | 0 | 3 | 0 | 0

9. Secondary Outcome: Number of Participants With Any SAEs
Description: as for outcome 6
Time Frame: Throughout the study period (Day 1 to Month 6)
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6
Participants | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Any AESIs
Description: as for outcome 7
Time Frame: Throughout the study period (Day 1 to Month 6)
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 18 | 6 | 18 | 6 | 18 | 6 | 18 | 18 | 6
Participants | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

11. Secondary Outcome: Geometric Mean Titers (GMT) of Neutralizing Titers Against Pseudovirus Bearing S Protein From Vaccine Encoded SARS-CoV-2 and Wild Type (WT) Strains
Description: The analyzed neutralizing titers were SARS-CoV-2 Neutralizing Titer BA.5 and SARS-CoV-2 Neutralizing Titer D614G. D= Day; M= Month.
Time Frame: At Days 1, 15 and 31, and at Month 6
Population: Analysis was performed on Per Protocol Set (PPS) which included participants who received investigational products, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination, who have neutralizing titer values against pseudovirus bearing S protein data, and without major protocol deviations. Only participants with data available at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Part A: Placebo Combined: Participants received placebo dose administered on Day 1. As described in the analysis plan, participants in the Part A, Group 1: Placebo, Part A, Group 2: Placebo, Part A and Group 3: Placebo were pooled for immunogenicity analyses.
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 3: mRNA CR-04 100 µg | Part A: Placebo Combined | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 16 | 17 | 17 | 18 | 18 | 18 | 5
Titers
  BA.5, D1 | 550.72 [325.81 to 930.89] | 526.95 [325.54 to 852.97] | 504.01 [287.71 to 882.94] | 320.87 [154.81 to 665.05] | 689.36 [402.31 to 1181.24] | 574.02 [385.58 to 854.56] | 493.05 [92.19 to 2636.84]
  BA.5, D15: number analyzed (Participants) | 16 | 17 | 17 | 18 | 18 | 17 | 5
  BA.5, D15 | 4271.90 [2751.76 to 6631.81] | 4720.61 [3082.55 to 7229.14] | 4795.20 [3132.57 to 7340.29] | 453.93 [298.47 to 690.36] | 2423.54 [1796.47 to 3269.50] | 3596.47 [2644.67 to 4890.81] | 589.81 [334.04 to 1041.42]
  BA.5, D31: number analyzed (Participants) | 14 | 17 | 16 | 18 | 17 | 17 | 5
  BA.5, D31 | 4197.66 [2747.44 to 6413.36] | 3607.13 [2463.89 to 5280.84] | 6591.72 [4448.81 to 9766.85] | 420.37 [288.08 to 613.40] | 2157.80 [1472.28 to 3162.53] | 2847.07 [1944.62 to 4168.31] | 602.35 [297.53 to 1219.45]
  BA.5, M6: number analyzed (Participants) | 11 | 13 | 15 | 15 | 18 | 12 | 5
  BA.5, M6 | 1414.22 [786.90 to 2541.66] | 1354.49 [793.70 to 2311.51] | 1919.56 [1164.60 to 3163.94] | 444.43 [266.94 to 739.93] | 1547.09 [1100.15 to 2175.61] | 1677.07 [1103.28 to 2549.28] | 540.16 [281.43 to 1036.75]
  D614G, D1 | 2502.06 [1839.63 to 3403.03] | 1409.21 [931.99 to 2130.80] | 1820.75 [1080.88 to 3067.05] | 1421.87 [706.04 to 2863.44] | 2139.66 [1353.70 to 3381.96] | 1604.51 [1013.28 to 2540.73] | 1702.33 [571.67 to 5069.18]
  D614G, D15: number analyzed (Participants) | 16 | 17 | 17 | 18 | 18 | 17 | 5
  D614G, D15 | 8073.12 [5651.68 to 11532.03] | 9990.27 [7096.52 to 14064.02] | 14543.96 [10348.31 to 20440.70] | 1654.35 [1186.60 to 2306.48] | 4661.13 [3673.40 to 5914.45] | 6363.85 [4982.55 to 8128.08] | 2129.10 [1358.56 to 3336.68]
  D614G, D31: number analyzed (Participants) | 14 | 17 | 16 | 18 | 17 | 17 | 5
  D614G, D31 | 6251.22 [4450.68 to 8780.17] | 7726.20 [5712.62 to 10449.51] | 12351.27 [9068.09 to 16823.16] | 1585.37 [1182.26 to 2125.92] | 4633.14 [3382.40 to 6346.37] | 7601.57 [5553.99 to 10404.02] | 2819.98 [1583.73 to 5021.26]
  D614G, M6: number analyzed (Participants) | 11 | 13 | 15 | 15 | 18 | 12 | 5
  D614G, M6 | 3813.02 [2511.62 to 5788.74] | 3970.88 [2713.92 to 5810.01] | 4645.04 [3267.21 to 6603.92] | 2441.97 [1715.51 to 3476.06] | 4059.06 [3244.67 to 5077.85] | 3342.96 [2541.75 to 4396.73] | 2571.87 [1680.53 to 3935.97]

12. Secondary Outcome: Geometric Mean Ratio (GMR) of Neutralizing Titers Against Pseudovirus Bearing S Protein From Vaccine Encoded SARS-CoV-2 and WT Strains
Description: as for outcome 11
Time Frame: At Days 15 and 31, and at Month 6 (compared with baseline [Day 1])
Population: Analysis was performed on PPS. Only participants with data available at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 3: mRNA CR-04 100 µg | Part A: Placebo Combined | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 16 | 17 | 17 | 18 | 18 | 17 | 5
Ratio
  BA.5, D15 | 9.25 [5.96 to 14.36] | 10.22 [6.68 to 15.66] | 10.38 [6.78 to 15.90] | 0.98 [0.65 to 1.50] | 3.91 [2.90 to 5.27] | 5.80 [4.27 to 7.89] | 0.95 [0.54 to 1.68]
  BA.5, D31: number analyzed (Participants) | 14 | 17 | 16 | 18 | 17 | 17 | 5
  BA.5, D31 | 8.57 [5.61 to 13.10] | 7.37 [5.03 to 10.78] | 13.46 [9.08 to 19.94] | 0.86 [0.59 to 1.25] | 3.43 [2.34 to 5.03] | 4.53 [3.09 to 6.63] | 0.96 [0.47 to 1.94]
  BA.5, M6: number analyzed (Participants) | 11 | 13 | 15 | 15 | 18 | 12 | 5
  BA.5, M6 | 2.76 [1.53 to 4.95] | 2.64 [1.55 to 4.51] | 3.74 [2.27 to 6.17] | 0.87 [0.52 to 1.44] | 2.26 [1.61 to 3.17] | 2.45 [1.61 to 3.72] | 0.79 [0.41 to 1.51]
  D614G, D15 | 4.68 [3.28 to 6.69] | 5.80 [4.12 to 8.16] | 8.44 [6.00 to 11.86] | 0.96 [0.69 to 1.34] | 2.53 [1.99 to 3.21] | 3.45 [2.70 to 4.41] | 1.15 [0.74 to 1.81]
  D614G, D31: number analyzed (Participants) | 14 | 17 | 16 | 18 | 17 | 17 | 5
  D614G, D31 | 3.50 [2.49 to 4.91] | 4.32 [3.20 to 5.85] | 6.91 [5.07 to 9.41] | 0.89 [0.66 to 1.19] | 2.43 [1.77 to 3.32] | 3.98 [2.91 to 5.45] | 1.48 [0.83 to 2.63]
  D614G, M6: number analyzed (Participants) | 11 | 13 | 15 | 15 | 18 | 12 | 5
  D614G, M6 | 1.99 [1.31 to 3.03] | 2.08 [1.42 to 3.04] | 2.43 [1.71 to 3.45] | 1.28 [0.90 to 1.82] | 2.01 [1.61 to 2.51] | 1.65 [1.26 to 2.18] | 1.27 [0.83 to 1.95]

13. Secondary Outcome: Number of Participants With Vaccine Response Rate (VRR) Based on Neutralizing Titers Against Vaccine Encoded SARS-CoV-2 and WT Strains
Description: VRR is expressed as the number of participants with a vaccine response, defined as at least a 4-fold greater neutralizing titer as compared to the titer at Day 1. D= Day; M= Month.
Time Frame: At Days 15 and 31, and at Month 6 (compared with baseline [Day 1])
Population: Analysis was performed on PPS. Only participants with data available at specified timepoints were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 3: mRNA CR-04 100 µg | Part A: Placebo Combined | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
Number analyzed (Participants) | 16 | 17 | 17 | 18 | 18 | 17 | 5
Participants
  BA.5, D15 | 11 | 13 | 14 | 2 | 7 | 13 | 0
  BA.5, D31: number analyzed (Participants) | 14 | 17 | 16 | 18 | 17 | 17 | 5
  BA.5, D31 | 12 | 12 | 15 | 0 | 5 | 11 | 0
  BA.5, M6: number analyzed (Participants) | 11 | 13 | 15 | 15 | 18 | 12 | 5
  BA.5, M6 | 3 | 3 | 7 | 1 | 4 | 3 | 0
  D614G, D15 | 6 | 8 | 12 | 0 | 3 | 9 | 0
  D614G, D31: number analyzed (Participants) | 14 | 17 | 16 | 18 | 17 | 17 | 5
  D614G, D31 | 5 | 8 | 11 | 0 | 4 | 8 | 0
  D614G, M6: number analyzed (Participants) | 11 | 13 | 15 | 15 | 18 | 12 | 5
  D614G, M6 | 2 | 3 | 4 | 2 | 2 | 3 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs: Day 1 to Day 7; Unsolicited AEs: Day 1 to Day 30. SAEs, MAAEs, AESIs: Day 1 up to study end (6 months post-investigational products administration).
Arm/Group | Part A, Group 1: mRNA CR-04 10 µg | Part A, Group 1: Placebo | Part A, Group 2: mRNA CR-04 30 µg | Part A, Group 2: Placebo | Part A, Group 3: mRNA CR-04 100 µg | Part A, Group 3: Placebo | Part B: mRNA CR-04 3 µg | Part B: mRNA CR-04 10 µg | Part B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6 | 0/18 | 0/6 | 0/18 | 0/6 | 0/18 | 0/18 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/6 | 1/18 | 0/6 | 0/18 | 0/6 | 0/18 | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 12/18 | 2/6 | 15/18 | 3/6 | 16/18 | 4/6 | 16/18 | 10/18 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: mRNA CR-04 10 µg (N=18) | Part A, Group 1: Placebo (N=6) | Part A, Group 2: mRNA CR-04 30 µg (N=18) | Part A, Group 2: Placebo (N=6) | Part A, Group 3: mRNA CR-04 100 µg (N=18) | Part A, Group 3: Placebo (N=6) | Part B: mRNA CR-04 3 µg (N=18) | Part B: mRNA CR-04 10 µg (N=18) | Part B: Placebo (N=6)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: mRNA CR-04 10 µg (N=18) | Part A, Group 1: Placebo (N=6) | Part A, Group 2: mRNA CR-04 30 µg (N=18) | Part A, Group 2: Placebo (N=6) | Part A, Group 3: mRNA CR-04 100 µg (N=18) | Part A, Group 3: Placebo (N=6) | Part B: mRNA CR-04 3 µg (N=18) | Part B: mRNA CR-04 10 µg (N=18) | Part B: Placebo (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 8 (8) | 1 (1) | 7 (7) | 1 (1) | 8 (8) | 2 (2) | 7 (7) | 5 (5) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 8 (8) | 0 (0) | 10 (10) | 1 (1) | 15 (15) | 0 (0) | 9 (9) | 6 (6) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
SARS-CoV-2 antibody test positive (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4) | 2 (2) | 11 (11) | 0 (0) | 6 (6) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 1 (1) | 4 (4) | 1 (1) | 8 (8) | 2 (2) | 7 (8) | 4 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Binge drinking (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT05972993/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT05972993/SAP_001.pdf